CLINICAL TRIAL: NCT02826616
Title: Chinese People's Liberation Army General Hospital
Brief Title: Effect of Trimetazidine During the Primary PCI on Cardiac Function in Patients With ST-elevation Myocardial Infarction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Qian geng, Chinese People's Liberation Army General Hospital, Chinese PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1672sdd
Record Dates: First submitted 2016-07-05; First posted 2016-07-11 (Estimated); Last update posted 2016-07-11 (Estimated); Status verified 2016-07

CONDITIONS: Cardiovascular Diseases
Keywords: Trimetazidine; ST-segment elevation myocardial; Reperfusion injury; Percutaneous coronary intervention
MeSH Terms: conditions — Cardiovascular Diseases; Reperfusion Injury | interventions — Trimetazidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Trimetazidine group (Experimental): Trimetazidine 60 mg 30 min before PCI and 20 mg for 12 months after surgery
  Interventions: Drug: Trimetazidine
- The control group (No Intervention): placebo 60 mg 30 min before PCI and 20 mg for 12 months after surgery

INTERVENTIONS:
Drug: Trimetazidine — Trimetazidine 60 mg 30min before PCI and 20 mg for 12 months after surgery
  Arms: Trimetazidine group

SUMMARY:
Giving preoperative loading dose of 60mg of trimetazidine can safely and effectively reduce the PCI-related myocardial damage for the patients undergoing selective PCI. but the effect of Trimetazidine during the primary PCI on cardiac function in patients with ST-elevation myocardial infarction is not sure. this study aim to study the effect of Trimetazidine during the primary PCI on cardiac function in patients with ST-elevation myocardial infarction.

DETAILED DESCRIPTION:
Investigators will enroll 240 patients with STEMI who were admitted to the Chinese PLA General Hospital between Januay 2017 and August 2017. STEMI was defined as typical chest pain lasting 30 min within the previous 12 h, a clear ST-segment elevation of N0.1 mV in ≥2 contiguous electrocardiographic leads, and elevated blood levels of troponin T. We randomly assign eligible patients in a 1:1 ratio to either 60mg of trimetazidine or oral placebo befor PCI. Trimetazidine group will accept 20mg of trimetazidine for 12 months after PCI and active Comparator will be given placebo for 12 months after PCI.

Primary end point of the study was the area of viable myocardium coming from MR delayed enhancement scan and main cardiovascular events concluding recurrent myocardial infarction, cardiac death, recurrent angina, acute heart failure. Secondary end point of the study was the change of LVEF. All adverse clinical events as well as study end points were monitored and adjudicated by the independent event committee. Each patient was contacted in every week after administration of the contrast, investigated main cardiovascular events (myocardial infarction,acute heart failure and death), and record any adverse events.

ELIGIBILITY:
Inclusion Criteria:

* STEMI patients: typical chest pain lasting 30 min within the previous 12 h, a clear ST-segment elevation of N0.1 mV in ≥2 contiguous electrocardiographic leads, and elevated blood levels of troponin T
* patients were scheduled to undergo diagnostic cardiac angiography or percutaneous coronary interventions

Exclusion Criteria:

* The combined use of trimetazidine contraindications;
* had cardiogenic shock,
* had a history of myocardial infarction, stent thrombosis, or renal insufficiency;
* had previously undergone coronary artery bypass surgery.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2016-07; Primary Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
TIMI flow grade | immediately post procedure
Myocardial infarct size according to MR delayed enhancement scan | 3 to 5 days after PCI
main cardiovascular events | follow up in one year

SECONDARY OUTCOMES:
change of the LVEF | follow up in one year

CONTACTS AND LOCATIONS:
Overall Officials: Dai Yun Chen, MD, Study Chair — Chinese PLA General Hospital
Locations (1):
- Chinese People's Liberation Army General Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Li J, Li X, Wang Q, Hu S, Wang Y, Masoudi FA, Spertus JA, Krumholz HM, Jiang L; China PEACE Collaborative Group. ST-segment elevation myocardial infarction in China from 2001 to 2011 (the China PEACE-Retrospective Acute Myocardial Infarction Study): a retrospective analysis of hospital data. Lancet. 2015 Jan 31;385(9966):441-51. doi: 10.1016/S0140-6736(14)60921-1. Epub 2014 Jun 23. PMID 24969506
- [Background] Lopaschuk GD, Ussher JR, Folmes CD, Jaswal JS, Stanley WC. Myocardial fatty acid metabolism in health and disease. Physiol Rev. 2010 Jan;90(1):207-58. doi: 10.1152/physrev.00015.2009. PMID 20086077
- [Background] Kantor PF, Lucien A, Kozak R, Lopaschuk GD. The antianginal drug trimetazidine shifts cardiac energy metabolism from fatty acid oxidation to glucose oxidation by inhibiting mitochondrial long-chain 3-ketoacyl coenzyme A thiolase. Circ Res. 2000 Mar 17;86(5):580-8. doi: 10.1161/01.res.86.5.580. PMID 10720420
- [Background] El Banani H, Bernard M, Baetz D, Cabanes E, Cozzone P, Lucien A, Feuvray D. Changes in intracellular sodium and pH during ischaemia-reperfusion are attenuated by trimetazidine. Comparison between low- and zero-flow ischaemia. Cardiovasc Res. 2000 Sep;47(4):688-96. doi: 10.1016/s0008-6363(00)00136-x. PMID 10974217
- [Background] Chen J, Zhou S, Jin J, Tian F, Han Y, Wang J, Liu J, Chen Y. Chronic treatment with trimetazidine after discharge reduces the incidence of restenosis in patients who received coronary stent implantation: a 1-year prospective follow-up study. Int J Cardiol. 2014 Jul 1;174(3):634-9. doi: 10.1016/j.ijcard.2014.04.168. Epub 2014 Apr 21. PMID 24809921
- [Background] Bonello L, Sbragia P, Amabile N, Com O, Pierre SV, Levy S, Paganelli F. Protective effect of an acute oral loading dose of trimetazidine on myocardial injury following percutaneous coronary intervention. Heart. 2007 Jun;93(6):703-7. doi: 10.1136/hrt.2006.107524. Epub 2007 May 8. PMID 17488771
- [Background] Kim JS, Kim CH, Chun KJ, Kim JH, Park YH, Kim J, Choi JH, Lee SH, Kim EJ, Yu DG, Ahn EY, Jeong MH. Effects of trimetazidine in patients with acute myocardial infarction: data from the Korean Acute Myocardial Infarction Registry. Clin Res Cardiol. 2013 Dec;102(12):915-22. doi: 10.1007/s00392-013-0611-0. Epub 2013 Aug 28. PMID 23982468
- [Background] El-Kady T, El-Sabban K, Gabaly M, Sabry A, Abdel-Hady S. Effects of trimetazidine on myocardial perfusion and the contractile response of chronically dysfunctional myocardium in ischemic cardiomyopathy: a 24-month study. Am J Cardiovasc Drugs. 2005;5(4):271-8. doi: 10.2165/00129784-200505040-00006. PMID 15984909
- [Background] Di Napoli P, Di Giovanni P, Gaeta MA, Taccardi AA, Barsotti A. Trimetazidine and reduction in mortality and hospitalization in patients with ischemic dilated cardiomyopathy: a post hoc analysis of the Villa Pini d'Abruzzo Trimetazidine Trial. J Cardiovasc Pharmacol. 2007 Nov;50(5):585-9. doi: 10.1097/FJC.0b013e31814fa9cb. PMID 18030070
- [Background] Gao D, Ning N, Niu X, Hao G, Meng Z. Trimetazidine: a meta-analysis of randomised controlled trials in heart failure. Heart. 2011 Feb;97(4):278-86. doi: 10.1136/hrt.2010.208751. Epub 2010 Dec 5. PMID 21134903
- [Background] Guler N, Eryonucu B, Gunes A, Guntekin U, Tuncer M, Ozbek H. Effects of trimetazidine on submaximal exercise test in patients with acute myocardial infarction. Cardiovasc Drugs Ther. 2003 Jul;17(4):371-4. doi: 10.1023/a:1027376529708. PMID 14696632
- [Background] Belardinelli R, Lacalaprice F, Faccenda E, Volpe L. Trimetazidine potentiates the effects of exercise training in patients with ischemic cardiomyopathy referred for cardiac rehabilitation. Eur J Cardiovasc Prev Rehabil. 2008 Oct;15(5):533-40. doi: 10.1097/HJR.0b013e328304feec. PMID 18797405
- [Background] Banach M, Rysz J, Goch A, Mikhailidis DP, Rosano GM. The role of trimetazidine after acute myocardial infarction. Curr Vasc Pharmacol. 2008 Oct;6(4):282-91. doi: 10.2174/157016108785909788. PMID 18855716
- [Background] Jogiya R, Kozerke S, Morton G, De Silva K, Redwood S, Perera D, Nagel E, Plein S. Validation of dynamic 3-dimensional whole heart magnetic resonance myocardial perfusion imaging against fractional flow reserve for the detection of significant coronary artery disease. J Am Coll Cardiol. 2012 Aug 21;60(8):756-65. doi: 10.1016/j.jacc.2012.02.075. Epub 2012 Jul 18. PMID 22818072
- [Derived] Qian G, A X, Jiang X, Jiang Z, Li T, Dong W, Guo J, Chen Y. Early Trimetazidine Therapy in Patients Undergoing Primary Percutaneous Coronary Intervention for ST Segment Elevation Myocardial Infarction Reduces Myocardial Infarction Size. Cardiovasc Drugs Ther. 2023 Jun;37(3):497-506. doi: 10.1007/s10557-021-07259-y. Epub 2021 Nov 12. PMID 34767131